CLINICAL TRIAL: NCT01369472
Title: A Randomized, Open-label, Single Dose, Dose-rising 10-sequence, 3-period Balanced Incomplete Blocked Clinical Trial to Evaluate Dose-proportionality of Dilatrend SR in Healthy Male Volunteers
Brief Title: Evaluating Dose-proportionality of Dilatrend Suspended-Release Capsule
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Collaborators: Asan Medical Center (Other)
Responsible Party: Jin Kim / Director, Clincal Research Department
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 125HPS11E
Record Dates: First submitted 2011-04-21; First posted 2011-06-09 (Estimated); Last update posted 2012-02-15 (Estimated); Status verified 2012-02

CONDITIONS: Chronic Stable Angina
MeSH Terms: conditions — Angina, Stable

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Dilatrend SR capsule 8mg (Experimental)
  Interventions: Drug: Dilatrend SR capsule
- Dilatrend SR capsule 16mg (Experimental)
  Interventions: Drug: Dilatrend SR capsule
- Dilatrend SR capsule 32mg (Experimental)
  Interventions: Drug: Dilatrend SR capsule
- Dilatrend SR capsule 64mg (Experimental)
  Interventions: Drug: Dilatrend SR capsule
- Dilatrend SR capsule 128mg (Experimental)
  Interventions: Drug: Dilatrend SR capsule

INTERVENTIONS:
Drug: Dilatrend SR capsule — single oral administration in period 1 or 2, 3 for each sequential group.

SUMMARY:
This study is designed to evaluate dose-proportionality of Dilatrend SR 8mg, 16mg, 32mg, 64mg, 128mg in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Age range 20 to 54 years, Body mass index of ≥19 and ≤26 healthy male volunteers
2. Able to participate in all procedure
3. SBP 90-140 mmHg, DBP 60-90 mmHg, Pulse rate 55-95 times/min
4. Have given written informed consent

Exclusion Criteria:

1. Have history of significant cardiovascular, hepatic, renal, pulmonary, hematologic, gastrointestinal, endocrine, musculoskeletal neurologic disease
2. Have history of gastrointestinal disease(Crohn's disease, gastrointestinal ulcer) or surgery(except for Appendectomy, Hernia)
3. Have allergy or hypersensitivity to carvedilol or any component of the formulation(aspirin, antibiotics)
4. Have history of drug abuse. A positive test for any drug(amphetamine, barbiturates, cocaine, opiates, benzodiazepines, THC, methadone, ect.) included in the urine drug screen.
5. Have herbal drug within 30days prior to the first IP administration, have ETC within 14days prior to the first IP administration, have OTC 7days prior to the first IP administration.
6. Have diet which may influence on the absorption, distribution, metabolism or excretion of drug(s), (Drinking over 1L of grapefruit juice within 7days prior to the first IP administration)
7. Have received an investigational drug within 60 days prior to the first IP administration
8. Have donated whole blood within 60 days prior or donation plasma within 30 days prior to the first IP administration
9. Have any metabolic enzyme including or inhibiting drugs like barbiturates within 30 days prior to the first IP administration.
10. A heavy caffeine/alcohol consumer or a heavy smoker(caffeine > 5 units/days. alcohol >21 units/week (1 unit=pure alcohol 10mL), Cigarette > 10 Cigarettes/day) or alcohol abuse.
11. Positive for Hepatitis B, Hepatitis C, HIV or syphilis

Ages: 20 Years to 54 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Dose-proportionality | 0(predose), 1, 2, 4, 5, 6, 8, 12, 16, 24, 36 and 48h
  AUClast
Dose-proportionality | 0(predose), 1, 2, 4, 5, 6, 8, 12, 16, 24, 36 and 48h
  AUC0-∞
Dose-proportionality | 0(predose), 1, 2, 4, 5, 6, 8, 12, 16, 24, 36 and 48h
  Cmax
Dose-proportionality | 0(predose), 1, 2, 4, 5, 6, 8, 12, 16, 24, 36 and 48h
  Tmax
Dose-proportionality | 0(predose), 1, 2, 4, 5, 6, 8, 12, 16, 24, 36 and 48h
  t½β

SECONDARY OUTCOMES:
Safety | 0(predose), 4, 8, 12, 24, 36, 48h and follow-up visit(22d±1d)
  Adverse Event/Serious Adverse Event monitoring Physical Examination, Vital Sign, 12-lead ECG, Lab Tests

CONTACTS AND LOCATIONS:
Overall Officials: KS Bae, Ph.D, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medcial Center, Songpa-gu, Seoul, South Korea